CLINICAL TRIAL: NCT07402174
Title: EIT- Guided Lung Recruitment in Pediatric Acute Respiratory Distress Syndrome
Brief Title: EIT- Guided Lung Recruitment in pARDS
Acronym: REMAV-EIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Giovanna Chidini, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1170_2021
Record Dates: First submitted 2025-06-11; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; EIT; Children
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Masking Description: This is a physiological, exploratory study involving real-time monitoring of ventilation using electrical impedance tomography (EIT). Masking is not applicable because the intervention, namely EIT-guided lung recruitment, requires direct observation and real-time adjustment by clinicians based on EIT data. Therefore, no participants, care providers, investigators, or outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EIT-Guided Recruitment (Experimental): This arm includes all participants undergoing a standardized staircase lung recruitment maneuver under continuous monitoring with Electrical Impedance Tomography (EIT). EIT is used to assess regional ventilation distribution and guide the titration of PEEP. Mechanical ventilation settings are adjusted based on individual EIT-derived responses. Respiratory mechanics, including transpulmonary pressure and compliance partitioning, are also recorded to evaluate physiological effects of recruitment.
  Interventions: Device: Electrical Impedance Tomography (EIT)-Guided Lung Recruitment

INTERVENTIONS:
Device: Electrical Impedance Tomography (EIT)-Guided Lung Recruitment — Staircase Recruitment Maneuver

SUMMARY:
Study Title:

EIT-Guided Lung Recruitment Maneuvers in Pediatric ARDS: Effects on Ventilation Distribution and Respiratory Mechanics

Study Objective:

The primary goal of this clinical trial is to determine whether lung recruitment maneuvers guided by Electrical Impedance Tomography (EIT) result in a more homogeneous ventilation distribution and less injurious ventilation in children with pediatric Acute Respiratory Distress Syndrome (pARDS). The study will assess changes in intrapulmonary gas distribution and respiratory mechanics during recruitment maneuvers using both EIT and partitioned respiratory mechanics.

This is a prospective cohort study involving children diagnosed with pARDS. Eligible participants will be consecutively enrolled over time and will undergo a standardized series of staircase lung recruitment maneuvers under continuous EIT monitoring. The final mechanical ventilation (MV) settings will be individualized and titrated based on the EIT-derived response to recruitment.

Main Research Questions:

How can lung recruitment maneuvers be performed safely in children with pARDS? How can we monitor the physiological effects of recruitment on respiratory mechanics? How does recruitment influence the distribution of ventilation within the lungs?

Eligible participants will undergo a series of staircase lung recruitment maneuvers under continuous EIT monitoring. The final mechanical ventilation (MV) settings will be titrated and individualized based on the EIT-derived response to recruitment.

DETAILED DESCRIPTION:
This is a prospective, single-center, interventional physiological study aiming to assess the effects of EIT-guided lung recruitment maneuvers on ventilation distribution and respiratory mechanics in children with pediatric acute respiratory distress syndrome (pARDS).

A total of 8 mechanically ventilated children diagnosed with moderate-to-severe pARDS will be enrolled within 48 hours from intubation. All patients will undergo a standardized staircase recruitment maneuver under continuous monitoring with Electrical Impedance Tomography (EIT). EIT will be used to assess regional ventilation distribution and guide the titration of PEEP to minimize lung collapse and overdistension. Partitioned respiratory mechanics will be measured through esophageal pressure monitoring to assess changes in lung and chest wall compliance, as well as transpulmonary pressure.

Primary outcome is the change in global inhomogeneity index (GI Index) measured before and after recruitment. Secondary outcomes include center of ventilation (CoV), regional ventilation delay (RVD).

Will also considerd overdistension and collapse percentages, changes in lung/chest wall mechanics.

This pilot study will provide physiological data to inform the design of future randomized trials on EIT-guided mechanical ventilation strategies in pediatric ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 month and 10 years
* Diagnosis of pediatric Acute Respiratory Distress Syndrome (pARDS) according to PALICC-2 criteria
* Invasive mechanical ventilation for less than 48 hours at the time of enrollment

Exclusion Criteria:

* Evidence or history of barotrauma (e.g., pneumothorax, pneumomediastinum)
* Presence of congenital heart disease with hemodynamic significance
* Known or suspected intracranial hypertension
* Presence of an implantable cardioverter-defibrillator (ICD)
* Parental o legal guardian refuse

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Global Inhomogeneity Index (GI) | Baseline (pre-intervention/procedure/surgery) Immediately after the intervention/procedure/surgery
  The Global Inhomogeneity Index (GI) is an EIT-derived quantitative measure of ventilation distribution heterogeneity across the lungs. A lower GI index indicates more homogeneous ventilation. GI will be calculated before and after the EIT-guided recruitment maneuver to assess the effect on regional ventilation distribution.

SECONDARY OUTCOMES:
Differences in Tidal Impedence | Baseline (pre-intervention/procedure/surgery) Immediately after the intervention/procedure/surgery
  Tidal impedance is a parameter derived from electrical impedance tomography (EIT) that reflects the regional distribution of ventilation during a tidal breath. Changes in electrical impedance measured between end-expiration and end-inspiration are proportional to changes in lung air volume, allowing real-time, bedside assessment of ventilation distribution.
Centre of Ventilation (CoV) | Baseline (pre-intervention/procedure/surgery) Immediately after the intervention/procedure/surgery
  The centre of ventilation is a quantitative measure that describes the geometric mean location of tidal ventilation within the lung along a predefined axis, most commonly the ventral-dorsal or cranio-caudal axis.
Changes in Regional Ventilation Delay (RVD) Index | Baseline (pre-intervention/procedure/surgery) Immediately after the intervention/procedure/surgery
  The RVD index quantifies the delay in regional ventilation during tidal breathing, indicating the degree of tidal recruitment or delayed filling. It reflects regional mechanical heterogeneity and is expected to decrease after effective lung recruitment.

OTHER OUTCOMES:
Partitioned Respiratory Mechanics | Baseline (pre-intervention/procedure/surgery) Immediately after the intervention/procedure/surgery
  Chest wall and lung elastance, measured by esophageal pressure monitorin

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Chidini, MD, Principal Investigator — Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico
Locations (2):
- Italy (2):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy
  - Fondazione Irccs Cà Granda Ospedale Maggiore Policlinico, Milan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including respiratory mechanics and EIT-derived ventilation metrics, will be made available to qualified researchers upon reasonable request. Data will be shared after publication of the primary results and following approval by the principal investigator and ethics committee.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication; available for up to 2 years.
Access Criteria: Researchers must submit a methodologically sound proposal and obtain approval from the principal investigator. In accordance with institutional policy, a formal Data Transfer Agreement (DTA) approved by the hospital's research foundation will be required before any data can be shared.
URL: https://www.policlinico.mi.it

REFERENCES:
- [Background] Frerichs I, Schiffmann H, Hahn G, Hellige G. Non-invasive radiation-free monitoring of regional lung ventilation in critically ill infants. Intensive Care Med. 2001 Aug;27(8):1385-94. doi: 10.1007/s001340101021. PMID 11511953
- [Background] Ren H, Xie L, Wang Z, Tang X, Ning B, Teng T, Qian J, Wang Y, Fu L, Zhao Z, Xiang L. Comparison of Global and Regional Compliance-Guided Positive End-Expiratory Pressure Titration on Regional Lung Ventilation in Moderate-to-Severe Pediatric Acute Respiratory Distress Syndrome. Front Med (Lausanne). 2022 May 23;9:805680. doi: 10.3389/fmed.2022.805680. PMID: 35677825; PMCID: PMC9167956.
- [Background] Cabezudo Ballesteros S, Sanabria Carretero P, Reinoso Barbero F. Review of electrical impedance tomography in the pediatric patient. Rev Esp Anestesiol Reanim (Engl Ed). 2024 Jun-Jul;71(6):479-485. doi: 10.1016/j.redare.2024.03.007. Epub 2024 Mar 6. PMID: 38458492.
- [Background] Soltész L, Leyens J, Vogel M, Muders T, Putensen C, Kipfmueller F, Dresbach T, Mueller A, Schroeder L. EIT guided evaluation of regional ventilation distributions in neonatal and pediatric ARDS: a prospective feasibility study. Respir Res. 2025 Feb 19;26(1):60. doi: 10.1186/s12931-025-03134-8. Erratum in: Respir Res. 2025 Jun 4;26(1):208. doi: 10.1186/s12931-025-03292-9. PMID: 39972380; PMCID: PMC11841312.
- [Background] Clasen D, Winter I, Rietzler S, Wolf GK. Changes in ventilation distribution during general anesthesia measured with EIT in mechanically ventilated small children. BMC Anesthesiol. 2023 Apr 12;23(1):118. doi: 10.1186/s12871-023-02079-z. PMID: 37046213; PMCID: PMC10091533.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT07402174/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT07402174/ICF_001.pdf